CLINICAL TRIAL: NCT07147517
Title: PREVENT: Preparedness Through Respiratory Virus Epidemiology and Community Engagement
Brief Title: Preparedness Through Respiratory Virus Epidemiology and Community Engagement
Acronym: PREVENT
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: San Ysidro Health Center (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Louise Laurent, MD/PhD, Principal Investigator, University of California, San Diego
Other Study IDs: 812427
Record Dates: First submitted 2025-08-14; First posted 2025-08-29 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Infection Virus; COVID -19; RSV; FLU
Keywords: respiratory pathogen testing; vending machine; implementation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Community Testing (A0): Component A0 participants (Community testing) will be members of the community who are interested in accessing testing for respiratory infections and will be asked to provide information that will then be used for screening for study Components A and/or B.
  Interventions: Other: Component A0
- Ongoing Testing (A): Participants in Component A (Ongoing Testing ) will undergo weekly symptom screening. If they report symptoms, they will be asked to provide a nasal swab and complete illness questionnaires on the day they report symptoms (Day 0) and again on Days 7 and 14.
  Interventions: Other: Component A1
- Immunology (A2): Participants in Component A Sub-study (Immunology) will provide blood and saliva/nasal fluid samples twice a year, as well as before and after infection and/or immunization against priority pathogens.
  Interventions: Other: Component A2
- Household Transmission (B): Participants in Component B (Household Transmission) will complete daily symptom questionnaires and nasal swabs for 14 days following enrollment, regardless of symptoms. Those who are symptomatic at enrollment will also complete retrospective daily diaries from symptom onset to the enrollment date. Additionally, they provide blood and/or saliva/nasal fluid samples at enrollment and again 28 days later.
  Interventions: Other: Component B

INTERVENTIONS:
Other: Component A0 — It will be implemented as a recruitment strategy. This strategy will enable members of the community to access no cost testing for respiratory infections. If a participant feels sick or thinks they have been exposed to a respiratory infection and wants to be tested, they can complete a symptoms and exposure survey in the PREVENT APP, retrieve a PCR test kit from a vending machine using a unique code received through the PREVENT APP, self-collect an anterior nares nasal swab following instructions provided, and return the test kit at one of the vending machines or drop off locations for the EXCITE lab to pick up and process. The anterior nares nasal swab will be tested for SARS-CoV-2, influenza, Respiratory Syncytial Virus, and other germs (viruses or bacteria) that cause respiratory infections. At the time of consent and registration for the Community Testing Component, participants will be used to screen for Cohorts A/B.
  Groups: Community Testing (A0)
Other: Component A1 — Participants will be invited to 'test' out the PREVENT App and a provide a 'baseline' sample to ensure competency for requesting a nasal swab, retrieving the test kit from a vending machine, self-collecting a sample, and returning the test for PCR testing, with the assistance of study staff. Weekly Symptom Surveys, Annual Surveys, and immunization status.
  Groups: Ongoing Testing (A)
Other: Component A2 — Investigators will collect immunologic specimens from a subset of participants in Component A (the subset herein referred to as Component A immunologic sub-study). Investigators will combine testing data from these immunologic specimens with multiple data elements already captured in Component A (such as data from pathogen testing and sequencing, survey data, medical records, or immunization services) and Component B (serum obtained at enrollment and 28 post-enrollment) to meet sub-study objectives. Overall, the Component A sub-study will provide critical insight into the immune response to respiratory pathogen infections and immunizations.
  Groups: Immunology (A2)
Other: Component B — Participants will be asked to complete the enrollment survey after enrolling in Component B if the survey has not already been completed as part of Component A. They will also be asked to complete:
  1. Daily anterior nares nasal swab collection
  2. All household participants, including the index case, will be asked to self-collect an enrollment swab and daily nasal swab specimens for 14 days and return them for testing.
  3. Mucosal specimen collection
  4. Survey data collection
  Groups: Household Transmission (B)

SUMMARY:
The CHARM network will be established through three primary institutions-Beth Israel Deaconess Medical Center (BIDMC), the University of California San Diego (UCSD), and the University of Washington (UW)-along with their subcontracting institutions. At UCSD and partner sites, the CHARM network will be implemented via the PREVENT project. All PREVENT participants will be consented in to Component A0 (Community Testing) and a subset of A0 participants will be invited to participate and will be consented into the other components: Component A (Ongoing Testing); Component A Sub-study (Immunology); Component B (Household Transmission).

Component A0 participants (Community testing) will be members of the community who are interested in accessing testing for respiratory infections and will be asked to provide limited information that will then be used for screening for study Components A and/or B.

Participants in Component A (Ongoing Testing ) will undergo weekly symptom screening. If they report symptoms, they will be asked to provide a nasal swab and complete illness questionnaires on the day they report symptoms (Day 0) and again on Days 7 and 14. Participants in Component A Sub-study (Immunology) will provide blood and saliva/nasal fluid samples twice a year, as well as before and after infection and/or immunization against priority pathogens.

Participants in Component B (Household Transmission) will complete daily symptom questionnaires and nasal swabs for 14 days following enrollment, regardless of symptoms. Those who are symptomatic at enrollment will also complete retrospective daily diaries from symptom onset to the enrollment date. Additionally, they provide blood and/or saliva/nasal fluid samples at enrollment and again 28 days later.

For all Components, UCSD will provide PCR test results for SARS-CoV-2, Influenza A/B, and RSV for nasal swab samples.

ELIGIBILITY:
Community Testing Component:

Inclusion:

- All community members are able to participate in the community testing component.

Exclusion:

- There is no exclusion criteria and participants will not be excluded based on pregnancy status or age.

For Component A:

Inclusion:

* All ages
* AND Lives in service area of a recruitment center (i.e., within range of courier pick up)
* AND Plans to remain living in a recruitment area for the next 2 years.

Exclusion:

* Inability to communicate in a language in which consent forms, materials, etc. are available
* OR Incarcerated
* OR Living in a congregate setting (e.g., assisted living, nursing home, university dormitories with shared bathroom and communal eating facilities)
* OR Unable/unwilling to participate in planned data and specimen collections
* OR Unable to comply with study procedures, as determined by study investigators
* OR Participation in clinical trials of investigational agents for respiratory viral infections during the three months prior to enrollment and for the duration of the study.

For Component B:

Inclusion:

Index case:

* Detection of priority respiratory pathogen via laboratory or point-of-care test on the day of eligibility screening or in the previous 5 days, AND
* Lives in service area of a recruitment center (i.e., within range of courier pick up), AND
* Lives in a household with ≥1 other person and plans to remain in the household for at least the duration of specimen collection (i.e., 14 days), AND
* Has not been hospitalized since the date of symptom onset.

Household contacts:

* Routinely sleep in the same household as index case and slept in household ≥1 night in the 7 days before index case symptom onset, AND
* Plan to remain in the household for at least the duration of specimen collection (i.e., 14 days).

Household:

* There is ≥1 non-ill household member (i.e., asymptomatic and has not tested positive for the virus of the index case) on the day of eligibility screening or in the previous 5 days,
* AND all symptomatic persons in the household had a symptom or diagnosis onset date on the day of eligibility screening or in the previous 5 days.

Exclusion:

Index case:

* Lives in a congregate setting (e.g., assisted living, nursing home, university dormitories with shared bathroom and communal eating facilities)
* Meet any A1 exclusion criteria

Household contacts:

* Has been hospitalized any time since date of primary case symptom onset
* Meets any A1 exclusion criteria

Household:

* The enrollment visit occurs >6 days after the first symptom onset of primary case
* The primary case in the household is not enrolled
* The primary case has been hospitalized any time after the date of symptom onset

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Investigators will include a large portion of San Diego County, which resides in HHS Region 9 and is the Southwestern-most county in the continental U.S, abutting the U.S./Mexico border.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Burden and Incident of respiratory illness via infection rates & questionnaires | 5 years
  Estimate the burden and incidence of respiratory illness in a community-based cohort of children and adults. A primary objective is to estimate the annual incidence of laboratory-confirmed symptomatic infection for primary respiratory viruses of interest (e.g., SARS-CoV-2, influenza A/B, and RSV A/B) stratified by age group (6 months-4 years, 5-17 years, 18-64 years, 65 or more years). The sample size and precision analysis assumes that the annual incidence of symptomatic laboratory-confirmed infections for priority respiratory viruses will range from 2% to 20%. Based on these assumptions, investigators plan to recruit 1,500 participants per age group. For each age group, sample size is calculated to provide a 95% confidence interval for the estimated annual incidence of symptomatic laboratory-confirmed infection with a precision ranging from ±0.5% to ±2% of the point estimate. This precision is contingent on the assumed annual incidence within the specified range (2% to 20%).
Implementation Effectiveness Questionnaire & Interviews | 5 years
  Assess implementation and effectiveness of interventions for respiratory pathogens. Investigators will describe the use of preventive behaviors, vaccination, and use of pharmaceutical interventions among the study participants. Investigators will explore associations between return of test result and preventive behaviors, healthcare seeking, and treatment via qualitative interviews and surveys.
Secondary Infection Rates | 5 years
  Estimate the secondary infection rates of respiratory pathogens in households and evaluate the effect of household, household member characteristics, and behaviors on household transmission. Sites will aim to recruit between 100 and 150 households per site, for a total of 450 households across the network. Assuming an average household size of 5 persons, research staff would recruit 450 index cases and 1800 household contacts.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UC San Diego, La Jolla, California
  - San Ysidro Health, San Ysidro, California

IPD SHARING:
Plan to Share IPD: Yes
Limited datasets with HIPAA data restricted to date of birth, date of study activities, and residence at the level of ZIP code/census tract will be shared with the study sponsor (CDC) and other investigators in the CHARM network, through a joint MTA/DUA and shared study Protocol and Dana Management Plan.